CLINICAL TRIAL: NCT01776541
Title: A Phase II, Randomized, Observer-Blind,Multi-Center, Study to Evaluate Safety, Tolerability and Immunogenicity of an Adjuvanted Cell Culture-Derived H5N1 Subunit Influenza Virus Vaccine at Two Different Formulations in Healthy Adult Subjects.
Brief Title: Safety and Immunogenicity of Two Doses of H5N1 Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V89_04
Record Dates: First submitted 2013-01-20; First posted 2013-01-28 (Estimated); Results first posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Pandemic H5N1 Influenza
Keywords: Influenza, Pandemic, H5N1, Adults
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- aH5N1c-High Dose (Experimental): Subjects received 2 injections of a high dose of cell culture-derived adjuvanted monovalent inactivated subunit H5N1 vaccine three weeks apart.
  Interventions: Biological: Adjuvanted H5N1 pandemic influenza vaccine
- aH5N1c-Low dose (Experimental): Subjects received 2 injections of a low dose of cell culture-derived adjuvanted monovalent inactivated subunit H5N1 vaccine three weeks apart.
  Interventions: Biological: Adjuvanted H5N1 pandemic influenza vaccine

INTERVENTIONS:
Biological: Adjuvanted H5N1 pandemic influenza vaccine — Comparison of two doses of aH5N1c vaccine

SUMMARY:
Evaluate Safety, Tolerability and Immune Response of Adjuvanted H5N1 Cell Culture Derived Influenza Vaccine in Adult Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects 18 to 64 years of age,
2. Individuals willing to provide written informed consent,
3. Individuals in good health,
4. Individuals willing to allow for their serum samples to be stored beyond the study period.

Exclusion Criteria:

1. Individuals not able to understand and follow study procedures,
2. History of any significant illness,
3. History of any chronic medical condition or progressive disease,
4. Presence of medically significant cancer,
5. Known or suspected impairment/alteration of immune function,
6. Presence of any progressive or severe neurologic disorder,
7. Presence of any bleeding disorders or conditions that prolongs bleeding time,
8. History of allergy to vaccine components,
9. Receipt of any other investigational product within 30 days prior to entry into the study,
10. History of previous H5N1 vaccination,
11. Receipt of any other type of seasonal vaccination within 2 months prior to entry into the study,
12. Receipt of any other vaccine within 2 weeks prior to entry into the study
13. Body temperature ≥38°C.0 (≥100.4° F) and/or acute illness within 3 days of intended study vaccination,
14. Pregnant or breast feeding,
15. Females of childbearing potential refusing to use acceptable method of birth control,
16. Body mass index (BMI) ≥ 35 kg/m2,
17. History of drug or alcohol abuse,
18. Any planned surgery during study period,
19. Individuals conducting the study and their immediate family members,
20. Individuals with behavioral or cognitive impairment or psychiatric diseases.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 979 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (8):
- United States (4):
  - 1 Miami Research Associates, Miami, Florida
  - 2 Mercy Health Research, St Louis, Missouri
  - 3 Saint Louis University, St Louis, Missouri
  - 4 Benchmark Medical Research, Austin, Texas
- Australia (3):
  - 48 Hunter Clinical Research, Newcastle, New South Wales
  - 46 CMAX, Adelaide, South Australia
  - 47 Linear Clinical Research, Nedlands, Western Australia
- 80 Faculty of Tropical Medicine, Bangkok, Thailand

REFERENCES:
- [Derived] Frey SE, Shakib S, Chanthavanich P, Richmond P, Smith T, Tantawichien T, Kittel C, Jaehnig P, Mojares Z, Verma B, Kanesa-Thasan N, Hohenboken M. Safety and Immunogenicity of MF59-Adjuvanted Cell Culture-Derived A/H5N1 Subunit Influenza Virus Vaccine: Dose-Finding Clinical Trials in Adults and the Elderly. Open Forum Infect Dis. 2019 Mar 1;6(4):ofz107. doi: 10.1093/ofid/ofz107. eCollection 2019 Apr. PMID 30968056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 4 centers in the US, 3 centers in Australia and 1 center in Thailand.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- High Dose: Subjects received 2 injections of a high dose of cell culture-derived adjuvanted monovalent inactivated subunit H5N1 vaccine three weeks apart.
- Low Dose: Subjects received 2 injections of a low dose of cell culture-derived adjuvanted monovalent inactivated subunit H5N1 vaccine three weeks apart.
Period: Overall Study
Arm/Group | High Dose | Low Dose
Started | 488 | 491
Completed | 432 | 416
Not Completed | 56 | 75
Not completed — Administrative Reason | 6 | 2
Not completed — Death | 4 | 0
Not completed — Lost to Follow-up | 27 | 48
Not completed — Unclassified | 5 | 4
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 12 | 20

BASELINE CHARACTERISTICS:
Groups:
- High Dose: Subjects received 2 injections of a high dose MF59 adjuvanted cell-culture derived monovalent H5N1 vaccine three weeks apart.
- Low Dose: Subjects received 2 injections of a low dose MF59 adjuvanted cell-culture derived monovalent H5N1 vaccine three weeks apart.
- Total: Total of all reporting groups
Arm/Group | High Dose | Low Dose | Total
Number analyzed (Participants) | 488 | 491 | 979
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (13.7) | 38.4 (14.2) | 38.7 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285 | 259 | 544
  Male | 203 | 232 | 435

OUTCOME MEASURES:

1. Primary Outcome: Percentages Of Subjects Achieving Hemagglutinin Inhibition (HI) Titers ≥40 Against A/H5N1 Strain.
Description: The optimal aH5N1c vaccine formulation was evaluated in terms of percentages of subjects achieving HI titers ≥40 against homologous A/H5N1 strain, three weeks after second vaccination with either low dose or high dose of aH5N1c vaccine, according to the Center for Biologics Evaluation and Research (CBER) criterion.
  CBER criterion for the adult population is met if the lower limit of the two-sided 95% confidence interval (CI) for the percentages of subjects achieving HI titer ≥40 meets or exceeds 70%.
Time Frame: Three weeks after 2nd vaccination (day 43)
Population: Analysis was done on the Full Analysis Set (FAS) i.e., the subjects who actually receive at least one dose of study vaccination and provide at least one evaluable serum sample both before (baseline) and after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 478 | 483
Percentages of subjects
  Day 1 | 4 [3 to 6] | 4 [2 to 6]
  Day 43 (N=451,440) | 85 [81 to 88] | 63 [58 to 68]

2. Primary Outcome: Percentages Of Subjects Achieving Seroconversion Against A/H5N1 Strain.
Description: Immunogenicity was measured in terms of the percentages of subjects achieving seroconversion or significant increase in HI titer against the vaccine strain, three weeks after receiving two injections of low dose or high dose of aH5N1c vaccine according to the CBER criterion.
  Seroconversion is defined as either a) in subjects with a prevaccination HI titer <10, a postvaccination titer ≥40; or b) in subjects with prevaccination HI titer ≥10, a minimum four-fold rise in postvaccination HI antibody titer.
  CBER criterion for the adult population is met if the lower limit of the two-sided 95% CI for the percentages of subjects achieving seroconversion for HI antibody titer meets or exceeds 40%.
Time Frame: Three weeks after 2nd vaccination (day 43)
Population: This analysis was done on the FAS population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 451 | 440
Percentages of subjects | 83 [79 to 86] | 61 [56 to 66]

3. Primary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events (AE), After Any Vaccination.
Description: Safety was assessed using the number of subjects who reported solicited local and systemic AEs following vaccination with either low or high dose of aH5N1c vaccine.
Time Frame: From day 1 through day 7 after any vaccination.
Population: Analysis was done on the safety dataset, i.e. the subjects in the exposed population who provided postvaccination safety data.
Measure: Number; unit: Number of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 473 | 471
Number of subjects
  Any Local | 322 | 236
  Injection site Erythema(N=471,471) | 4 | 0
  Injection site Induration(N=471,471) | 54 | 35
  Injection site Ecchymosis(N=472,471) | 9 | 6
  Injection site Pain(N=471,470) | 318 | 235
  Any Systemic | 223 | 209
  Nausea(N=472,471) | 54 | 48
  Myalgia(N=472,469) | 108 | 78
  Arthralgia(N=471,467) | 70 | 52
  Headache(N=471,469) | 126 | 114
  Fatigue(N=471,469) | 125 | 108
  Loss of Appetite(N=472,469) | 53 | 38
  Malaise(N=472,467) | 117 | 97
  Fever (≥38°C)(N=472,469) | 11 | 9
  Treatment of pain and (or) fever(N=471,470) | 40 | 31
  Prevention of pain and (or) fever(N=471,470) | 7 | 14
  Fever (≥40°C)(N=472,469) | 1 | 0

4. Primary Outcome: Number of Subjects Reporting Unsolicited AEs After Any Vaccination.
Description: Safety was assessed using the number of subjects who reported any unsolicited adverse events, adverse events possibly or probably related to study vaccine, serious adverse events (SAEs), new onset of chronic diseases (NOCDs), medically attended AEs, AEs of special interest (AESIs), AEs leading to withdrawal from study following vaccination with either low or high dose of aH5N1c vaccine.
Time Frame: Any unsolicited AEs - day 1 through day 22 after any vaccination. SAEs, NOCDs. medically attended AEs, AESIs, AEs leading to study withdrawal- day 1 to day 387
Population: as for outcome 3
Measure: Number; unit: Number of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 476 | 475
Number of subjects
  Any AEs | 94 | 92
  At least possibly related AEs | 39 | 31
  Any SAEs | 20 | 8
  Deaths | 4 | 0
  Medically attended AEs | 171 | 153
  AEs resulting in premature withdrawal from study | 4 | 0
  AEs of Special Interest | 1 | 0
  AEs leading to New Onset of Chronic Disease | 11 | 14

5. Secondary Outcome: Geometric Mean Ratios Against A/H5N1 Strain Following 2-dose Vaccination Schedule of Either Low Dose or High Dose aH5N1c Vaccine.
Description: Immunogenicity was measured as the geometric mean ratio (GMR). The ratio of postvaccination to prevaccination HI GMTs, 3 weeks after first vaccination, 3 weeks after second vaccination and 12 months after second vaccination of either low dose or high dose of aH5N1c is reported.
  The criterion is met according to the European Committee for Medicinal Products for Human Use (CHMP) criterion if the geometric mean increase GMR (day 43/day 1) in HI antibody titer is >2.5 for subjects 18-60 years of age.
Time Frame: Day 1; day 22; day 43 and day 387
Population: Analysis was done on the FAS set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 464 | 461
Ratio
  Day22/Day1 | 5.37 [4.6 to 6.27] | 2.43 [2.07 to 2.84]
  Day43/Day1 (N=451,440) | 41 [34 to 49] | 11 [8.68 to 13]
  Day387/Day1 (N=411,395) | 1.95 [1.73 to 2.19] | 1.24 [1.1 to 1.4]

6. Secondary Outcome: Percentages Of Subjects With HI Titers ≥40 Against A/H5N1 Strain.
Description: Immunogenicity was assessed in terms of percentage of subjects achieving HI titers ≥40, 3 weeks after first vaccination, 3 weeks after second vaccination and 12 months after second vaccination of either low dose or high dose of aH5N1c according to the CHMP criterion.
  European Licensure (CHMP) criterion is met if the percentage of subjects achieving (at day 43) HI titers ≥40 is >70%.
Time Frame: Day 1, day 22, day 43 and day 387
Population: Analysis was done on the FAS set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 478 | 483
Percentages of subjects
  Day 1 | 4 [3 to 6] | 4 [2 to 6]
  Day 22 (N=464,461) | 52 [47 to 56] | 30 [26 to 35]
  Day 43 (N=451,440) | 85 [81 to 88] | 63 [58 to 68]
  Day 387 (N=411,395) | 27 [22 to 31] | 11 [8 to 15]

7. Secondary Outcome: Percentages Of Subjects Achieving Seroconversion Against A/H5N1 Strain.
Description: Immunogenicity was assessed in terms of percentages of subjects achieving seroconversion in HI titers, 3 weeks after first vaccination, 3 weeks after second vaccination and 12 months after second vaccination of either low dose or high dose aH5N1c vaccine according to the CHMP criterion.
  Seroconversion is defined as: a) for subjects with a prevaccination HI titer <10, a postvaccination titer ≥40; or b) for subjects with prevaccination HI titer ≥10, a minimum four-fold rise in postvaccination HI antibody titer.
  The criterion is met according to the European (CHMP) guideline if the percentage of subjects achieving seroconversion (at day 43) is >40%.
Time Frame: Day 22, day 43 and day 387
Population: Analysis was done on the FAS set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 464 | 461
Percentages of subjects
  Day 22 | 48 [44 to 53] | 27 [23 to 31]
  Day 43 (N=451,440) | 83 [71 to 91] | 61 [45 to 75]
  Day 387 (N=411,395) | 22 [18 to 26] | 9 [6 to 12]

ADVERSE EVENTS:
Time Frame: Solicited local and systemic adverse events from day 1 to 7. SAEs and Unsolicited AEs (other than SAEs) from day 1 to 387.
Description: All Solicited AEs are classified as systematic assessment and all unsolicited AEs are classified as non-systematic assessment.
  Subjects who did not provide unsolicited safety data were excluded from safety evaluation.
Groups:
- Total: Total of high dose and low dose groups.
Arm/Group | High Dose | Low Dose | Total
Serious Adverse Events (participants affected / at risk) | 20/485 | 8/490 | 28/975
Other Adverse Events (participants affected / at risk) | 371/485 | 324/490 | 695/975
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=485) | Low Dose (N=490) | Total (N=975)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 1 | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 1 | 2
JAUNDICE (Hepatobiliary disorders) | 0 | 1 | 1
APPENDICITIS (Infections and infestations) | 1 | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0 | 1
INFLUENZA (Infections and infestations) | 1 | 0 | 1
PNEUMONIA (Infections and infestations) | 2 | 0 | 2
PYELONEPHRITIS (Infections and infestations) | 1 | 0 | 1
SEPSIS (Infections and infestations) | 2 | 0 | 2
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 1 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 1
LIMB CRUSHING INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 1
POST LAMINECTOMY SYNDROME (Injury, poisoning and procedural complications) | 0 | 1 | 1
POSTOPERATIVE ADHESION (Injury, poisoning and procedural complications) | 1 | 0 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 1
LARYNGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 1
NERVE COMPRESSION (Nervous system disorders) | 1 | 0 | 1
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 1
ABORTION MISSED (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 2
NEPHROLITHIASIS (Renal and urinary disorders) | 2 | 0 | 2
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
RAYNAUD'S PHENOMENON (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=485) | Low Dose (N=490) | Total (N=975)
NAUSEA (Gastrointestinal disorders) | 58 | 51 | 109
FATIGUE (General disorders) | 125 | 111 | 236
INJECTION SITE ERYTHEMA (General disorders) | 76 | 61 | 137
INJECTION SITE HAEMORRHAGE (General disorders) | 42 | 28 | 70
INJECTION SITE INDURATION (General disorders) | 59 | 41 | 100
INJECTION SITE PAIN (General disorders) | 319 | 244 | 563
MALAISE (General disorders) | 117 | 97 | 214
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 53 | 44 | 97
DECREASED APPETITE (Metabolism and nutrition disorders) | 56 | 38 | 94
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 75 | 60 | 135
MYALGIA (Musculoskeletal and connective tissue disorders) | 112 | 82 | 194
HEADACHE (Nervous system disorders) | 134 | 120 | 255

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No